CLINICAL TRIAL: NCT04112524
Title: Comparison of Quantitative Metamorphopsia- Measurements in Patients With mCNV
Status: Completed | Type: Observational
Sponsor: PD Dr. med. Katja Hatz (Other)
Responsible Party: Sponsor-Investigator, PD Dr. med. Katja Hatz, Head of clinical research and medical retina, Vista Klinik, Vista Klinik
Organization: Vista Klinik (Other)
Other Study IDs: Metamorphopsia Study
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Metamorphopsia
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients from routine treatment: all 30 patients from Routine Treatment, only observational
  Interventions: Device: App

INTERVENTIONS:
Device: App — * Alleye® Test Alleye® Test is a mobile medical software application indicated for the detection and characterization of metamorphopsia. For the mean Alleye score (±standard deviation (SD) deviations of dots from an ideal line are calculated for each eye.
  * AMD-A Metamorphopsia Detector® Is based on the Amsler grid. The software uses the concept of a negative image: a distorted image can be straightened by moving the mouse. Degree and dimension of distorted lines or scotoma are transformed into indices.

SUMMARY:
The myopic CNV (mCNV) is a blood vessel neoplasm starting from the choroid, based on pathological myopia (severe myopia).

Choroidal neovascularization secondary to pathological myopia is the most common cause of severe visual impairment in myopic patients younger than 50 years old. Because untreated small fibrovascular membranes cause rapid damage to the photoreceptors, timely treatment is required in view of poor spontaneous prognosis1.

Metamorphopsia is the first functional impairment which occurs in mCNV - visual acuity loss and scotoma follow later.

There is a need for better and quicker quantifying of the metamorphopsia in mCNV patients.

The aim of this study is to detect metamorphopsia and verify correlations of different indexes with disease activity or not, measured in Optical Cohorence Tomography (OCT), best corrected visual acuity (BCVA), Vision related quality of life questionnaire (NEI-VFY-25) and quantify severity of metamophopsia.

DETAILED DESCRIPTION:
The myopic CNV is a neovascularization starting from the choroid and growing into the space between choroid and retina, based on pathological myopia (severe myopia). Choroidal neovascularization secondary to pathological myopia (mCNV) is the most common cause of severe visual impairment in myopic patients younger than 50 years old.1 As untreated subretinal fibrovascular membranes cause rapid damage to the photoreceptors, timely treatment is required in view of poor spontaneous prognosis.1

Metamorphopsia is the first functional impairment which occurs in mCNV - visual acuity loss and scotoma follow later. The Amsler Grid, a qualitative paper test developed the swiss ophthalmologist Marc Amsler (1891 - 1968), is a square-shaped grid used to detect or monitor metamorphopsia or scotoma involving the central visual field in various disorders of the macula and optic nerve head11.

Myopic CNV patients use the Amsler Grid as a home monitoring device for qualitative detection of metamorphopsia by checking the grid regularly11. Due to subretinal scarring in mCNV interpretation is often difficult and early changes cannot be detected and quantified. Until now there are no quantitative measurements for mCNV monitoring in clinical use.

Recently, two devices to detect and monitor metamorphopsia using smart phones and PCs, respectively, have been developed for use in choroidal neovascularization in age-related macular degeneration.5,6

* Alleye® Test Alleye® Test is a mobile medical software application indicated for the detection and characterization of metamorphopsia. For the mean Alleye score (±standard deviation (SD) deviations of dots from an ideal line are calculated for each eye.5
* AMD-A Metamorphopsia Detector® Is based on the Amsler grid. The software uses the concept of a negative image: a distorted image can be straightened by moving the mouse. Degree and dimension of distorted lines or scotoma are transformed into indices.6

This study was designed to find out whether these metamorphopsia applications are suitable for patients with mCNV and to find out if mCNV patients can benefit for a quicker detecting of the metamorphopsia.

Therefore, the aim of this study is to detect metamorphopsia and verify correlations of different indexes with disease activity or not, measured in Optical Cohorence Tomography (OCT), best corrected visual Acuity (BCVA), Vision related quality of life questionnaire (NEI-VFY-25) and quantify severity of metamophopsia.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of mCNV involving the juxtafoveal or/and foveal region
* BCVA >0.1 (20/200, Snellen)
* ability to follow the study procedures
* given written consent to participation
* >18 years

Exclusion Criteria:

* history of vitreoretinal surgery (including membrane peeling and retinal detachment surgery) to the study eye
* presence of macula foramen or epiretinal membrane with significant distortion of retinal architecture
* history of any side effects to Tropicamide eye drops

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients in retina- routine control
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Metamorphopsia index change from baseline (no mCNV activity) to month 6 and 12 and all visits in between (disease activity dependent) for the following two devices - AMD-A Metamorphopsia Detector® (app4eyes - TEST) - Alleye® Test | 1 year
  Metamorphopsia index change (disease activity)

SECONDARY OUTCOMES:
CRT (central retinal thickness) measured in OCT | 1 year
  CRT change (disease activity)
-outer retina disruption score within central 1mm (measured in OCT) -maximum CNV thickness within central 1mm (measured in OCT) -area of pigment epithelium atrophy within central 1mm measured in autofluorescence imaging | 1 year
  Change of outer Retina disruption score and maximum CNV thickness
NEI VFQ-25 questionnaire -BCVA (best corrected visual acuity) | 1 year
  Change in BCVA

CONTACTS AND LOCATIONS:
Locations (1):
- Vista Klinik, Binningen, Basel-Landschaft, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
when we finished our study (master Thesis) and published (if possible), then we will participant our data